CLINICAL TRIAL: NCT04842435
Title: To Study the Efficacy, Safety and Pharmacokinetics of COVID-globulin, in Addition to Standard Therapy for the Treatment of Patients With a Moderate COVID-19 Form
Brief Title: Clinical Study in the Treatment of Patients With Moderate Course of COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Microgen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGK-P-II/III-00-003/2020
Record Dates: First submitted 2021-04-12; First posted 2021-04-13 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: COVID-19; Moderate COVID-19; Pharmacokinetic parameters
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Stage 1 study will enroll 156 subjects with moderate COVID-19 who will be randomized into the four groups.
  Stage 2 will include 220 subjects who will be divided into two groups.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Stage 1. Group 1 (Experimental): Group 1 - 39 subjects who will receive a single intravenous infusion of COVID-globulin at a dose of 1 mL/kg in addition to standard therapy
  Interventions: Drug: COVID-globulin
- Stage 1. Group 2 (Experimental): Group 2 - 39 subjects who will receive a single intravenous infusion of COVID-globulin at a dose of 2 mL/kg in addition to standard therapy
  Interventions: Drug: COVID-globulin
- Stage 1. Group 3 (Experimental): Group 3 - 39 subjects who will receive a single intravenous infusion of COVID-globulin at a dose of 4 mL/kg in addition to standard therapy
  Interventions: Drug: COVID-globulin
- Stage 1. Group 4 (Placebo Comparator): Group 4 - 39 subjects who will receive a single intravenous infusion of placebo at a dose of 1 mL/kg in addition to standard therapy
  Interventions: Drug: Placebo
- Stage 2. Group 1 (Active Comparator): Group 1 - 110 subjects who will receive a single intravenous infusion of COVID-globulin at a dose defined at Stage 1 in addition to standard therapy
  Interventions: Drug: COVID-globulin
- Stage 2. Group 2 (Placebo Comparator): Group 2 - 110 subjects who will receive a single intravenous infusion of placebo at a dose equal to the COVID-globulin dose in addition to standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COVID-globulin — In a Stage 1 study, COVID globulin is administered to clinical study subjects randomized to groups 1, 2, or 3 by intravenous drip in one of three doses of 1 mL/kg, 2 mL/kg, or 4 mL/kg The initial drug administration rate is from 0.01 mL/kg to 0.02 mL/kg of body weight per minute for 30 minutes. If the drug is well tolerated, the rate of administration can be gradually increased to a maximum of 0.12 mL/kg of body weight per minute. In order to control the drug administration rate, infusion shall be performed with an infusion pump.
  In a Stage 2 study, COVID globulin is administered to clinical study subjects randomized to group 1 by intravenous drip at a dose found optimal based on the results of Stage 1 study.
  Other Names: Anti-coronavirus human immunoglobulin
  Arms: Stage 1. Group 1; Stage 1. Group 2; Stage 1. Group 3; Stage 2. Group 1
Drug: Placebo — In a Stage 1 study, Placebo is administered to clinical study subjects randomized to groups 4 by intravenous drip at a dose of 1 mL/kg.
  The initial drug administration rate is from 0.01 mL/kg to 0.02 mL/kg of body weight per minute for 30 minutes. If the drug is well tolerated, the rate of administration can be gradually increased to a maximum of 0.12 mL/kg of body weight per minute. In order to control the drug administration rate, infusion shall be performed with an infusion pump.
  In a Stage 2 study, placebo is administered to clinical study subjects randomized to group 2 by intravenous drip at a dose equal to the study drug dose.
  Other Names: 0.9% NaCl solution
  Arms: Stage 1. Group 4; Stage 2. Group 2

SUMMARY:
Study of safety, efficacy and pharmacokinetics, dose selection

DETAILED DESCRIPTION:
Objective:

To study the efficacy, safety and pharmacokinetics of COVID-globulin, in addition to standard therapy for the treatment of patients with a moderate COVID-19 form.

Study Objectives:

The study comprises two stages, 1 and 2. Stage 1 tasks

1. to determine and compare the safety parameters of COVID-globulin after a single infusion at doses of 1 mL/kg, 2 mL/kg, 4 mL/kg and placebo in addition to standard therapy in the treatment of patients with COVID-19;
2. to determine and compare the efficacy parameters of COVID-globulin after a single infusion at doses of 1 mL/kg, 2 mL/kg, 4 mL/kg and placebo in addition to standard therapy in the treatment of patients with COVID-19;
3. to determine the optimal therapeutic dose of COVID-globulin for the treatment of patients with moderate COVID-19 by comparing the safety and efficacy parameters of doses of 1 mL/kg, 2 mL/kg, 4 mL/kg and placebo;
4. to study the pharmacokinetic parameters of COVID-globulin in the blood plasma of patients after a single infusion at a dose of 1 mL/kg, 2 mL/kg, 4 mL/kg, in addition to standard therapy for the treatment of patients with moderate COVID-19.

Stage 2 tasks

1. to study the efficacy of COVID-globulin in addition to standard therapy for the treatment of patients with moderate COVID-19;
2. to study the safety of COVID-globulin in addition to standard therapy for the treatment of patients with moderate COVID-19;
3. to conduct a comparative analysis of the efficacy and safety of a group of patients with moderate COVID-19 who receive COVID-globulin in addition to the standard therapy, and a group of patients who receive placebo in addition to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are able to sign the informed consent form to partic-ipate in the clinical study;
2. Patients of both sexes at the age of 18-65 years of age;
3. Positive SARS-CoV-2 RNA test result obtained by PCR during the current episode of COVID-19 disease;
4. One or more clinical manifestations of ARI (acute respiratory infection) or patient complaints: cough (dry or scanty sputum), edema (including during exercise), chest congestion, sore throat, nasal congestion, or mild rhinorrhea, impairment or loss of smell (hyposmia or anosmia), loss of taste (dysgeusia), conjunctivitis, weakness, muscle pain, headache, vomiting, diarrhea, skin manifestations).
5. Patients with a moderate course of COVID-19, determined on the basis of at least one of the criteria specified in the Interim Guide-lines of the Ministry of Health (assessed from the moment of mani-festation of the disease symptoms):

   * Body Т > 38 °C
   * RR > 22/min
   * SpO2 < 95 % (at the atmospheric air)
   * CRP of the blood serum > 10 mg/L
6. CT changes typical of viral lesions (minimal or moderate lesion vol-ume; CT 1-2, no more than 72 hours before screening)
7. Patients meeting the requirements of the Clinical Study Protocol;
8. Negative pregnancy test (for women with preserved reproductive potential).

Exclusion Criteria:

1. A history of allergic reactions to human blood products;
2. Allergic reactions to the components of the study drug;
3. Hypersensitivity to human immunoglobulin;
4. Positive direct Coombs test (antiglobulin test);
5. Condition requiring invasive oxygen support at Screening;
6. Subjects with mild, severe, extremely severe COVID-19, as well as those at an outpatient treatment and not scheduled for hospitali-zation;
7. Administration of blood products or blood derivatives within 3 months prior to enrollment;
8. Administration of any antiviral, immunomodulatory drugs after the manifestation of COVID-19 (except for those to be prescribed dur-ing the study / included in the standard therapy);
9. Pathology of the immune system (primary and secondary immu-nodeficiencies, deficiency of class A immunoglobulin (IgA) and / or the presence of IgA antibodies, autoimmune diseases);
10. Child Pugh class B and C liver cirrhosis;
11. Diabetes mellitus type 1.
12. Diseases of the thyroid gland with decompensation.
13. Signs of severe CNS lesions (past serious brain injury, meningitis, history of ischemic stroke, encephalopathy of various etiologies, epilepsy, etc.);
14. Serious blood diseases, current or in the history (for example, baseline anemia Hb < 80, myeloid leukemia, myelodysplastic syn-drome, etc.);
15. The period after the coronary artery bypass grafting / stenting of at least 3 months prior to enrollment;
16. Malignant neoplasm of any localization at present or within 5 years before enrollment into the study, except for completely healed carcinoma in situ;
17. Conditions and diseases, other than COVID-19, known from anam-nesis, accompanied by blood hypercoagulability syndrome and a trend for thrombosis (such as sickle cell anemia, polycythemia, hemostatic disorders);
18. Severe dyslipidemia in the history;
19. Disseminated intravascular coagulation syndrome, thrombosis and thromboembolism of any localization, known from the history;
20. CKD-EPI GFR < 30 mL/min at screening;
21. History of chronic III-IV FC heart failure;
22. Pregnancy or lactation;
23. Participation in any other clinical study within the last 3 months;
24. A history of tuberculosis, cancer or a positive reaction to HIV infec-tion, hepatitis B and C, syphilis according to the history;
25. Impossibility of intravenous administration of the drug;
26. Severe visual and/or hearing impairments, severe speech impair-ments and/or other abnormalities that may prevent the patient from adequate cooperation during the study);
27. Mental diseases in the history;
28. A history of alcohol, drug or medicinal product abuse;
29. Patients who, in the opinion of the investigator, are clearly or likely to be unable to understand and evaluate the information on this study within the informed consent signing process, in particular regarding the expected risks and possible discomfort;
30. Other diseases, symptoms or conditions not listed above that can be an obstacle to participation in a clinical study in the investiga-tor's opinion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects in the study groups in whom, during the first 7 days after drug administration, one of the following events developed according to the laboratory-instrumental methods or on the basis of a clinical presentation | 7 days
  Laboratory-instrumental methods or on the basis of a clinical presentation:
  * development of acute renal injury stage 2 or higher, assessed by the AKIN (Acute Kidney Injury Network) scale;
  * development of myocardial dysfunction or acute coronary pathology;
  * development of thrombolytic complications;
  * development of a cytokine storm;
  * development of an acute respiratory distress syndrome (ARDS);
  * an increase in the degree of lung lesion, as determined by the CT;
  * negative dynamics of CRP with an increase in the indicator by more than 30 % compared to the baseline value;
  * an increase in the D-dimer indicator by more than 2 times compared with the corresponding indicator at the time of hospitalization;
  * aggravation of clinical symptoms, as determined by the WHO Ordinal Scale, compared with the baseline value.
  (Aggravation refers to a decrease in a WHO score by 1 point or more as compared to the value at Visit 1)

SECONDARY OUTCOMES:
All-cause mortality | 28 days
  All-cause mortality (follow-up period of 28 days after the treatment initiation).
The elimination time of the SARS-CoV-2 virus | 11 days
  The elimination time of the SARS-CoV-2 virus from the upper respiratory tract (follow-up period of 11 days after the treatment initiation).
The median time to clinical improvement on the WHO Ordinal Scale for Clinical Improvement | 28 days
  The median time to clinical improvement on the WHO Ordinal Scale for Clinical Improvement (follow-up period of 28 days after the treatment initiation) using the Hazard Ratio score.
The incidence of severe and extremely severe COVID-19 disease | 28 days
  The incidence of severe and extremely severe COVID-19 disease (follow-up period of 28 days after the treatment initiation).
The need for respiratory support | 28 days
  The need for respiratory support (follow-up period of 28 days after the treatment initiation).
The need for invasive mechanical ventilation of the lungs, ECMO | 28 days
  The need for invasive mechanical ventilation of the lungs, ECMO (follow-up period of 28 days after the treatment initiation).
Time to cancellation of oxygen support | 28 days
  Time to cancellation of oxygen support, if any, days (follow-up period of 28 days after the treatment initiation).
The need to stay at the intensive care unit | 28 days
  The need to stay at the intensive care unit (follow-up period of 28 days after the treatment initiation).
Duration of fever (≥ 380C), days | 28 days
  Duration of fever (≥ 380C), days (follow-up period of 28 days after the treatment initiation).
The dynamics of the decrease in points on the NEWS scale | 11 days (max. 28 days)
  The dynamics of the decrease in points on the NEWS scale.
  NEWS uses six physiological measurements: respiratory rate; oxygen saturation; temperature; systolic blood pressure; heart rate and level of consciousness. Each scores 0-3 and individual scores are added together for an overall score. An additional one points are added if the patient is receiving oxygen therapy.
  Higher scores mean a worse outcome.
Dynamical CRP, ferritin, D-dimer values | 10 days
  Dynamical CRP, ferritin, D-dimer values.
  Local laboratories of research centers will be used for laboratory tests and assessments.
  After collecting and verification 100% values of laboratory parameters according to the Protocol from all local laboratories, the units of measurement will be unified before Statistical process control by valid formulas for transitions.
Changes in the degree of lung lesion determined by the CT | 7 days
  Changes in the degree of lung lesion determined by the CT (the result is assessed on the 7th day before the subject is discharged from the hospital compared to the baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Andreevna Bykova, Study Director — JSC "SIC "Microgen"
Locations (21):
- Russia (21):
  - 9. State Autonomous Healthcare Institution "Professor A. F. Agafonov Republican Clinical Infectious Hospital", Kazan'
  - 13. State Budgetary Healthcare Institution "Specialized Clinical Infectious Diseases Hospital" of the Ministry of Health of the Krasnodar Territory, Krasnodar
  - 6. State Budgetary Healthcare Institution "Scientific and Research Institute Professor S. V. Ochapovskiy Territorial Clinical Hospital" of the Ministry of Health of the Krasnodar Territory, Krasnodar
  - 1. State Budgetary Institution of Healthcare of Moscow "City Clinical Hospital No. 40 of the Moscow Department of Health", Moscow
  - 14. State Budgetary Institution of Healthcare of Moscow "Infectious Clinical Hospital No. 2" of the Moscow Department of Health, Moscow
  - 16. State Budgetary Institution of Healthcare of Moscow "Infectious Clinical Hospital No. 1" of the Moscow Department of Health, Moscow
  - 18. State Budgetary Institution of Healthcare of Moscow "City Clinical Hospital No. 52 of the Moscow Department of Health", Moscow
  - 19. State Budgetary Institution of Healthcare of Moscow "City Clinical Hospital of V.P. Demikhova of the Moscow Department of Health", Moscow
  - 20. State Budgetary Institution of Healthcare of Moscow "Scientific and Research Institute of N.V. Sklifosovskiy of the Moscow Department of Health", Moscow
  - 21. State Budgetary Institution of Healthcare of Moscow "City Clinical Hospital No. 4 of the Moscow Department of Health", Moscow
  - 3. State Budgetary Healthcare Institution of Moscow "City Clinical Hospital No. 24 of the Moscow Department of Health", Moscow
  - 7. Federal State Budgetary Institution "Central Clinical Hospital with an Outpatient Facility" of the Administrative Directorate of the President of the Russian Federation, Moscow
  - 4. Federal State Budgetary Educational Institution of Higher Education "Orenburg State Medical University" of the Ministry of Health of the Russian Federation, Orenburg
  - 10. Federal State Budgetary Educational Institution of Higher Education "Academician I. P. Pavlov Ryazan State Medical University" of the Ministry of Health of the Russian Federation, Ryazan
  - 5. Saint Petersburg State Budgetary Healthcare Institution "City Hospital No. 40 of the Kurortny Region", Saint Petersburg
  - 12. Federal State Budgetary Educational Institution of Higher Education "Samara State Medical University" of the Ministry of Health of the Russian Federation, Samara
  - 11. Regional State Budgetary Healthcare Institution "Clinical Hospital No. 1", Smolensk
  - 17. Federal State Budgetary Educational Institution of Higher Education "Bashkiria State Medical University" of the Ministry of Health of the Russian Federation, Ufa
  - 8. State Budgetary Healthcare Institution of the Yaroslavl Region "Yaroslavl Regional Clinical Hospital of War Veterans - International Center for Problems of the Elderly "Zdorovoye Dolgoletiye", Yaroslavl
  - 15. Municipal Autonomous Institution "Central City Clinical Hospital No. 24", Yekaterinburg
  - 2. State Budgetary Institution of Healthcare of the Moscow Region "Zhukovskiy City Clinical Hospital", Zhukovskiy

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date
Access Criteria: Anyone who wishes to access the data